CLINICAL TRIAL: NCT05084274
Title: Optimising Preconceptual Health in Subfertile PCOS Patients. Implementation of a Lifestyle Modification Program Before Fertility Treatment, Impact on Health Related Quality of Life and Obstetric Outcome
Brief Title: Optimising Preconceptual Health in Subfertile PCOS Patients Using a Lifestyle Modification Program
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Co-investigators have left and not been replaced.
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LSPCOLMMDV
Record Dates: First submitted 2021-10-06; First posted 2021-10-19 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-02

CONDITIONS: Infertility, Female; Polycystic Ovarian Syndrome; Lifestyle
MeSH Terms: conditions — Infertility, Female; Polycystic Ovary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle intervention group (Active Comparator): 12-week lifestyle modification programme through face-to-face lifestyle counseling and physiotherapy combined with a follow-up programme using video consultations and online training sessions
  Interventions: Behavioral: Lifestyle program
- Standard-of-care group (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Lifestyle program — If the patient is allocated to the interventional group, the lifestyle modification program will be planned/started immediately after the intake at the fertility clinic. The lifestyle modification program has a duration of 12 weeks in which the subject will receive follow-up by the endocrinologist/diabetologist and dietitian to re-ceive an active dietary intervention plan, follow-up by the physiotherapist where sessions to start with physical exercise will be given. Monthly follow-up visits with the coordinating PCOS-midwife will be planned to enhance the subject's knowledge about PCOS and give emotional support. At the moment of randomization, the PCOS coordinating midwife will immediately plan all necessary appointments, with the endocrinologist and dietitian, physiotherapist and PCOS-coordinator, for the 12-week lifestyle program. This way, patients will have a clear overview of the following 12 weeks.
  Arms: Lifestyle intervention group

SUMMARY:
Patients will be randomly assigned to a group where they undergo a 12-week lifestyle modification program prior to their fertility treatment, or a group where they are entitled to start their fertility treatment without prior lifestyle modification program.

DETAILED DESCRIPTION:
When allocated to the control arm patients will receive the standard of care combined with the foreseen questionnaires and bio-electric impedance analysis for body composition and ergospirometry. When the patient is allocated to the interventional arm she will receive a 12-week lifestyle modification program prior to her fertility treatment. The lifestyle modification program will consist of dietary advice, advice for physical activity and emotional support. After the 12-week program the fertilty treatment will start as per routine practice. Questionnaires, ergospirometry and bio-electric impedance analysis will also be performed at the foreseen moments.

ELIGIBILITY:
Inclusion Criteria:

* Subfertile patients between >18- <38 years old requesting fertility treatment at our centre
* PCOS phenotypes A, B, C and D according to the NIH 2012 extension of the ESHRE/ASRM 2003 diagnostic criteria
* BMI >27 and <38 (Jiskoot et al. 2017)
* Nulliparous women
* Patient gives consent voluntarily

Exclusion Criteria:

Patients will be excluded if they:

* do not meet the ESHRE/ASRM 2003 diagnostic PCOS criteria
* Have a BMI <27 and >38 (Jiskoot et al. 2017)
* Need Surgical sperm retrieval
* Use donor eggs
* Need Pre-implantation genetic testing (PGT)
* Multiparous women
* cannot reliably fill out the questionnaires or comprehend the intervention, because of a language barrier

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-02-26 (Actual)

PRIMARY OUTCOMES:
body weight | 12 weeks after start of intervention
  body weight (kg)
body composition | 12 weeks after start of intervention
  body composition (Total Body Fat and Fat Free Mass), measured by using bio-electric im-pedance analysis (BIA)

CONTACTS AND LOCATIONS:
Overall Officials: Michel De Vos, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No